CLINICAL TRIAL: NCT01593436
Title: The Effects of Mindfulness and RelaxationTraining for Insomnia (MRTI) on Postmenopausal Women: a Randomized Clinical Trial.
Brief Title: Mindfulness and RelaxationTraining for Insomnia (MRTI) on Postmenopausal Women: a Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, marcelo csermak garcia, principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0708/11
Record Dates: First submitted 2012-04-23; First posted 2012-05-08 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Primary Insomnia
Keywords: insomnia,menopause, polysomnography, mindfulness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Mindfulness; Meditation; Menopause

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mindfulness training (Active Comparator): mindfulness training for patients with insomnia
  Interventions: Behavioral: mindfulness training
- polysomnography and actigraphy (No Intervention): The intention is to assess the sleep architecture of meditators and non meditators women without menopausal insomnia by polysomnographic , actigraphy, and questionnaires to assess sleep quality and emotional state

INTERVENTIONS:
Behavioral: mindfulness training — mindfulness interventions for 8 weeks for a group of menopausal insomniacs
  Other Names: mindfulness,; meditation,; sleep pattern in meditators women in menopause
  Arms: mindfulness training

SUMMARY:
Summary

Introduction: Insomnia is a symptom of sleep disorders most prevalent. Primary insomnia, the investigators analyzed, often related to stress states acquired, generalized anxiety and stress, which are important factors that disrupt normal sleep. The investigators point out a fact that still intrigue the students of medicine and sleep that is distorted perception of sleep by the sleepless nights, polysomnography shows greater effectiveness than that perceived by them. On the other hand, there is evidence that mindfulness techniques may reduce symptoms of stress and anxiety as well as improve the general attention, which may contribute to a better perception of the effectiveness of sleep. In addition, there are studies showing that meditation is associated with metabolic and neurophysiological characteristics similar to normal sleep. Objectives: To compare sleepless menopausal women trained for 8 weeks in the technique of mindfulness insomniac postmenopausal untrained and also assess the quality of sleep experienced meditators menopausal comparing them to the group of healthy postmenopausal women untrained in the art.

DETAILED DESCRIPTION:
Groups will be assessed by actigraphy, polysomnography and questionnaires for assessing stress, depression, anxiety, quality of life, self-pity, subjective states such as sedation and other physical or mental attitudes, vitality, emotional state and attentiveness. Moreover, prospective memory participants will be evaluated by means of a task as close as possible to real life conditions of the volunteers (green) and also the working memory is assessed by a test called specific counting span. Menopausal women will be evaluated for the presence or absence of bruxism compared to ordinary meditators, all postmenopausal.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria for postmenopausal women with insomnia:

* be available to attend any training program of mindfulness (1 time per week for 8 weeks) and perform the suggested practices home.
* be available to perform the tests at home polysomnography (overnight) and other tests.
* Be available to perform the blood collection
* meet the criteria established in accordance with DSM-IV-TR for insomnia
* age 50 to 65 years.
* Women in menopause: women presenting with absence of menstruation in the past year and either FSH greater than 30.
* Have a BMI value lower than 30.
* Not having undergone any previous treatment against insomnia.
* Not having made use of hypnotics for at least 15 days.

Inclusion criteria for women without menopausal insomnia

* be available to perform the examinations polysomnographic (overnight) and other tests.
* To meditators, having trained as a practice of mindfulness meditation for at least 3 years 3 times a week.
* Age: 50 to 65 years
* Being a woman and being in menopause: women presenting failures or lack of regular menstrual periods last year.

Exclusion Criteria:Exclusion criteria for menopausal women with insomnia

* being under drug treatment, subjects will not be accepted that use of benzodiazepines, antihistamines, hypnotics, herbal sleeping pills, sedatives, antidepressants, antipsychotics, stimulants (amphetamine, caffeine, modafinil), corticosteroids, bronchodilators and beta blockers.
* being under psychological or psychiatric treatment.
* present history of neurological or psychiatric diseases such as severe psychotic disorders.
* having other sleep disorders like narcolepsy, sleep-disordered breathing, sleep apnea with an index greater than 15 / h, circadian rhythm disorder or parasomnias.
* 4 years of schooling below complete primary school

Exclusion criteria for menopausal women without complaints of insomnia:

* being under drug treatment, subjects will not be accepted that use of benzodiazepines, antihistamines, hypnotics, herbal sleeping pills, sedatives, antidepressants, antipsychotics, stimulants (amphetamine, caffeine, modafinil), corticosteroids, bronchodilators and beta blockers.
* being in psychological treatments.
* having had contact with a meditation technique.
* present history of neurological or psychiatric diseases such as severe psychotic disorders, as well as anxiety and depression.
* women presenting failures or regular period last year.
* 4 years of schooling below complete primary school
* submit any sleep disorders

Ages: 50 Years to 66 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The investigators intend to evaluate the effectiveness of mindfulness training in postmenopausal women with insomnia | two years
  The insomniacs were trained for 8 weeks in mindfullness,and they had a 30-minute meditation class once a week. They also received a meditation audio,to practice three times a day for 15 minutes in their homes.The control group was not infirm intervention. The meditation group showed relief of the symptoms of insomnia, indicated by Pittsburgh Insomnia Index, actigraphy and polysomnography, improving the overall quality of sleep and decreasing number of awakening.The control group remained with the same symptoms and complaints of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Helena hachul Campos, advisor, Study Director — UNIFESP-Federal University of Sao Paulo
Locations (1):
- Associacao Fundo de Incentivo a Psicofarmacologia Sao Paulo, SP, Brazil, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Garcia MC, Kozasa EH, Tufik S, Mello LEAM, Hachul H. The effects of mindfulness and relaxation training for insomnia (MRTI) on postmenopausal women: a pilot study. Menopause. 2018 Sep;25(9):992-1003. doi: 10.1097/GME.0000000000001118. PMID 29787483